CLINICAL TRIAL: NCT07399067
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Proof-of-Concept Study to Evaluate the Efficacy and Safety of IBI3002 in Patients With Moderate to Severe Atopic Dermatitis
Brief Title: A Proof-of-Concept Study of IBI3002 in Patients With Moderate to Severe Atopic Dermatitis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIBI3002B201
Record Dates: First submitted 2026-01-15; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- IBI3002 Dose Level 2 with Dosing Interval 1 (Experimental): Participants will receive IIBI3002 Dose Level 2subcutaneously according to the study schedule.
  Interventions: Drug: IBI3002
- Placebo (Placebo Comparator): Matched placebo will be administered subcutaneously according to the study schedule.
  Interventions: Drug: Placebo
- IBI3002 Dose Level 3 with Dosing Interval 1 (Experimental): Participants will receive IBI3002 Dose Level 3 subcutaneously according to the study schedule.
  Interventions: Drug: IBI3002
- IBI3002 Dose Level 1 with Dosing Interval 1 (Experimental): Participants will receive IBI3002 Dose Level 1subcutaneously according to the study schedule.
  Interventions: Drug: IBI3002
- IBI3002 Dose Level 1 with Dosing Interval 2 (Experimental): Participants will receive IBI3002 Dose Level 1 subcutaneously according to the study schedule.
  Interventions: Drug: IBI3002

INTERVENTIONS:
Drug: IBI3002 — IBI3002 will be administered subcutaneously at the assigned dose level and dosing interval.
  Arms: IBI3002 Dose Level 1 with Dosing Interval 1; IBI3002 Dose Level 1 with Dosing Interval 2; IBI3002 Dose Level 2 with Dosing Interval 1; IBI3002 Dose Level 3 with Dosing Interval 1
Drug: Placebo — Matched placebo will be administered subcutaneously at the same schedule as IBI3002.
  Arms: Placebo

SUMMARY:
The primary objective of this Phase 2 study is to evaluate the efficacy and safety of IBI3002 in patients with moderate to severe Atopic Dermatitis (AD).

DETAILED DESCRIPTION:
This is a Phase 2, multicenter, randomized, double-blind, placebo-controlled, parallel-group study designed to evaluate the efficacy, safety, tolerability, pharmacokinetics (PK), immunogenicity, and pharmacodynamic (PD) effects of IBI3002 in Chinese participants with moderate-to-severe AD.

A total of approximately 96 participants with moderate-to-severe AD are planned for enrollment. Baseline disease severity, categorized as moderate (vIGA-AD = 3) or severe (vIGA-AD = 4), will be used as a stratification factor. Eligible participants will be randomized to five treatment groups in a 2:1:1:2:2 ratio, including matched placebo and multiple dose levels of IBI3002 administered subcutaneously at specified intervals.

The study will assess changes in clinical efficacy measures, PK parameters, immunogenicity, and PD biomarkers over the treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and sign written informed consent prior to any study procedures and willingness to comply with study requirements throughout the study.
2. Age between 18 and 75 years old (inclusive).
3. Body weight ≥40 kg, with a Body Mass Index (BMI) between 18 and 35 kg/m² (inclusive).
4. Participants of childbearing potential and their partners must agree to strictly follow contraceptive measures specified in the protocol during the study and for 6 months after study completion.
5. At screening, participants must meet the Hannifin & Rajka diagnostic criteria, and have been diagnosed with AD for at least 12 months.
6. At screening and randomization, participants must have an EASI score ≥16, vIGA-AD score ≥3, involved body surface area (BSA) ≥10%, and baseline PP-NRS ≥4.
7. History of inadequate response to topical therapy within the past 12 months, or documented medical reasons making topical therapy unsuitable (e.g., severe adverse reactions or safety concerns).

Exclusion Criteria:

1. Clinically significant diseases that may affect safety or study participation, including but not limited to psychiatric, CNS, cardiovascular, digestive, respiratory, urinary, hematologic, or metabolic disorders.
2. Known history of active tuberculosis or clinically suspected tuberculosis (including but not limited to pulmonary tuberculosis, lymph node tuberculosis, tuberculous pleurisy, etc.); or chest imaging suggestive of suspected tuberculosis; or any other clinical evidence of latent tuberculosis.
3. History of malignant tumors, except for surgically removed or cured localized basal cell carcinoma (BCC) or squamous cell carcinoma (SCC) of the skin.
4. History of severe systemic allergic reactions (e.g., anaphylaxis, laryngeal edema).
5. Fainting at the sight of needles, blood, or inability to tolerate intravenous puncture.
6. Pregnant or breastfeeding women, or female participants who test positive for pregnancy during screening or at randomization.
7. Receipt of other investigational drugs within 3 months or 5 half-lives before randomization (whichever is longer), or current participation in another clinical trial.
8. Severe infection (defined as requiring hospitalization or intravenous anti-infective therapy) or trauma within 3 months before randomization; history of surgery within 3 months; infection requiring systemic treatment within 1 month; or planned surgical procedures during the study.
9. Receipt of any live vaccines (except influenza vaccine) within 1 month before randomization, or planning to receive vaccination during the study.
10. History of parasitic infections within 6 months before screening, or planning to travel to parasite-endemic countries/regions in Africa, South America, and southern parts of Asia (including Southeast Asia, India, Nepal) within 6 months after study completion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2027-03-23 (Estimated); Study Completion 2027-05-27 (Estimated)

PRIMARY OUTCOMES:
Percentage change from baseline in the Eczema Area and Severity Index (EASI) score at Week 16 | Week 16
  Percentage change from baseline in the EASI score at Week 16 in participants with moderate to severe AD after administration of IBI3002. EASI is used to assess the severity and extent of AD by evaluating four disease signs: (1) erythema, (2) induration/papulation, (3) excoriation, and (4) lichenification. The total EASI score ranges from 0 to 72, with higher scores indicating more severe disease.
  EASI-50: ≥ 50% reduction in score from baseline; EASI-75: ≥ 75% reduction in score from baseline; EASI-90: ≥ 90% reduction in score from baseline. EASI-100: 100% reduction in score from baseline.

SECONDARY OUTCOMES:
Number of participants with Adverse Events (AEs)/Serious Adverse Events (SAEs) | Up to 20 weeks
  Percentage of participants who have experienced AEs/SAEs.
Pharmacokinetic parameter Cmax of IBI3002 following multiple doses | Up to 20 weeks
  Maximum observed concentration (Cmax) of IBI3002 following multiple doses.
Pharmacokinetic parameter Tmax of IBI3002 following multiple doses | Up to 20 weeks
  Time to reach maximum concentration (Tmax) of IBI3002 following multiple doses.
Pharmacokinetic parameter AUC of IBI3002 following multiple doses | Up to 20 weeks
  Area under the concentration-time curve (AUC) of IBI3002 following multiple doses.
Immunogenicity of IBI3002 following multiple doses | Up to 20 weeks
  Immunogenicity will be assessed by the incidence of anti-drug antibodies (ADAs) in participants receiving IBI3002.
Percentage of participants with a validated Investigator's Global Assessment for Atopic Dermatitis (vIGA-AD) score of 0 (clear) or 1 (almost Clear) and a reduction ≥ 2 points from baseline at Week 16 | Week 16
  The vIGA-AD is a 5-point scale used to assess the overall severity of AD based on key acute clinical signs, including erythema, induration/papulation, oozing/crusting (lichenification excluded). The rating of clear (0), almost clear (1), mild (2), moderate (3) and severe (4), will be assessed at scheduled visits. The vIGA-AD must be conducted before the EASI assessment. The vIGA-AD is a static assessment performed independently of previous scores and is conducted prior to the EASI assessment.
Proportion of participants with a ≥ 50% improvement from baseline in EASI (EASI-50) at Week 16 | Week 16
  Proportion of patients with a ≥ 50% improvement from baseline in EASI (EASI-50) at Week 16. EASI is used to assess the severity and extent of AD by evaluating four disease signs: (1) erythema, (2) induration/papulation, (3) excoriation, and (4) lichenification. The total EASI score ranges from 0 to 72, with higher scores indicating more severe disease.
  EASI-50: ≥ 50% reduction in score from baseline; EASI-75: ≥ 75% reduction in score from baseline; EASI-90: ≥ 90% reduction in score from baseline. EASI-100: 100% reduction in score from baseline.
Proportion of participants with a ≥ 75% improvement from baseline in EASI (EASI-75) at Week 16 | Week 16
  Proportion of patients with a ≥ 75% improvement from baseline in EASI (EASI-75) at Week 16. EASI is used to assess the severity and extent of AD by evaluating four disease signs: (1) erythema, (2) induration/papulation, (3) excoriation, and (4) lichenification. The total EASI score ranges from 0 to 72, with higher scores indicating more severe disease.
  EASI-50: ≥ 50% reduction in score from baseline; EASI-75: ≥ 75% reduction in score from baseline; EASI-90: ≥ 90% reduction in score from baseline. EASI-100: 100% reduction in score from baseline.
Proportion of participants with a ≥ 90% improvement from baseline in EASI (EASI-90) at Week 16 | Week 16
  Proportion of patients with a ≥ 90% improvement from baseline in EASI (EASI-90) at Week 16. EASI is used to assess the severity and extent of AD by evaluating four disease signs: (1) erythema, (2) induration/papulation, (3) excoriation, and (4) lichenification. The total EASI score ranges from 0 to 72, with higher scores indicating more severe disease.
  EASI-50: ≥ 50% reduction in score from baseline; EASI-75: ≥ 75% reduction in score from baseline; EASI-90: ≥ 90% reduction in score from baseline. EASI-100: 100% reduction in score from baseline.
Proportion of participants with a 100% Improvement from baseline in EASI (EASI-100) at Week 16 | Week 16
  Proportion of patients with a 100% improvement from baseline in EASI (EASI-100) at Week 16. EASI is used to assess the severity and extent of AD by evaluating four disease signs: (1) erythema, (2) induration/papulation, (3) excoriation, and (4) lichenification. The total EASI score ranges from 0 to 72, with higher scores indicating more severe disease.
  EASI-50: ≥ 50% reduction in score from baseline; EASI-75: ≥ 75% reduction in score from baseline; EASI-90: ≥ 90% reduction in score from baseline. EASI-100: 100% reduction in score from baseline.
Proportion of participants achieving vIGA-AD 0 or 1 at Week 16 | Week 16
  The vIGA-AD is a 5-point scale assessing overall disease severity based on key acute clinical signs. Scores range from 0 (clear) to 4 (severe). The proportion of participants with a score of 0 (clear) or 1 (almost clear) will be assessed at Week 16.
Proportion of participants with ≥2-point reduction from baseline in vIGA-AD score at Week 16 | Week 16
  The vIGA-AD is a 5-point scale assessing overall disease severity based on key acute clinical signs. Scores range from 0 (clear) to 4 (severe). The proportion of participants achieving a ≥2-point reduction from baseline will be assessed at Week 16.
Proportion of participants with ≥4-point reduction from baseline in weekly average of daily Peak Pruritus Numerical Rating Scale (PP-NRS) during at Week 16 | Week 16
  The PP-NRS is a patient-reported tool used to assess the intensity of pruritus (itch) over a 24-hour recall period. Participants rate their worst itch on an 11-point scale from 0 (no itch) to 10 (worst itch imaginable) by answering: "On a scale of 0 to 10, how would you rate your worst itch during the previous 24 hours?" Higher scores indicate greater itch severity. At least 4 daily scores out of 7 days are required to calculate the weekly average score.

CONTACTS AND LOCATIONS:
Locations (1):
- China-japan Friendship Hospital, Beijing, Beijing Municipality, China